CLINICAL TRIAL: NCT02219620
Title: Examining the Effects of (MiM) Treatment on Emotional and Cognitive Functioning of Residents in Long-term Care
Acronym: MiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Holly Matto, Associate Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-953118
Record Dates: First submitted 2014-07-28; First posted 2014-08-19 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Emotion; Impaired Cognition
Keywords: creative arts; older adults; intervention study
MeSH Terms: conditions — Cognition Disorders | interventions — Movement; Social Control, Formal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music, Imagery, Movement intervention (Experimental): Music, Imagery, Movement intervention: psychosocial intervention incorporating Music, Imagery and Movement
  Interventions: Behavioral: Music, Imagery, Movement
- Social Control (Active Comparator): social control/interaction group
  Interventions: Behavioral: Social Control

INTERVENTIONS:
Behavioral: Music, Imagery, Movement — Implementation of music, art and imagery activation, and movement in group modality
  Arms: Music, Imagery, Movement intervention
Behavioral: Social Control — social conversational group facilitated by care counselor
  Arms: Social Control

SUMMARY:
To examine the effects of a music, imagery, and movement (MiM) intervention on emotional and cognitive functioning in residents living in a community-based adult long-term care facility.

Hypothesis 1: Residents who participate in the MiM group will improve in emotional functioning, as compared to residents in the control group.

Hypothesis 2: Residents who participate in the MiM group will improve in cognitive functioning, as compared to residents in the control group.

DETAILED DESCRIPTION:
To implement a community-based integrated music, art and imagery, and movement intervention to improve mood and promote cognitive functioning in older adult residents living in a long-term care facility.

ELIGIBILITY:
Inclusion Criteria:

* Resident in assisted living at long-term care facility with MMSE score above 20

Exclusion Criteria:

* co-morbid psychiatric diagnosis and/or staff clinical evaluation that determines inappropriateness for study inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
emotional functioning | pre-post 10 week treatment and 6 week FU

SECONDARY OUTCOMES:
cognitive functioning | pre-post 10 week intervention and 6 week FU

CONTACTS AND LOCATIONS:
Overall Officials: Holly Matto, Ph.D., Principal Investigator — George Mason University; Cathy Tompkins, Ph.D., Principal Investigator — George Mason University; Emily Ihara, Ph.D., Principal Investigator — George Mason University
Locations (1):
- Assisted Living at Birmingham Green, Manassas, Virginia, United States